CLINICAL TRIAL: NCT04060407
Title: Phase Ib/II Study Combining CD24Fc With Checkpoint Inhibitors for Patients With Metastatic Melanoma
Brief Title: CD24Fc With Ipilimumab and Nivolumab to Decrease irAE (CINDI)
Acronym: CINDI
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Oncoimmune, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Huntsman Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7110-004; R44CA250889 (NIH); CD24-004-CINDI (Other: OncoImmune)
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Advanced Melanoma (Experimental): Patients with advanced melanoma.
  Interventions: Drug: CD24Fc; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: CD24Fc — CD24Fc will be administrated as IV infusion in a dose of 480 mg, q3w x 4, then q4w for up to 6 times.
  Other Names: Human CD24 and human IgG Fc Fusion Protein
Drug: Ipilimumab — Ipilimumab will be administrated as IV infusion, q3w x 4. For metastatic melanoma, the dose will be 3mg/kg, q3w x4.
  Other Names: Yervoy, MDX-010.
Drug: Nivolumab — Nivolumab will be administrated as IV infusion. For metastatic melanoma, the dose will be 1mg/kg, q3w x 4, then 480 mg, q4w for up to 1 year.
  Other Names: Opdivo, MDX-1106, BMS-936558

SUMMARY:
This is a phase Ib/II clinical trial to test safety and efficacy of combining CD24Fc with ipilimumab and nivolumab to decrease irAE, with built-in interim analyses, and safety and response stopping rules.

DETAILED DESCRIPTION:
This is a phase 1b/II clinical trial using a fixed recommended phase 2 dose (RP2D) of CD24Fc to explore the safety and efficacy of combining CD24Fc with ipilimumab and nivolumab to reduce the toxicity of immunotherapy combination, in patients who are naïve to anti-PD1/L1 based checkpoint inhibitors. The dosing of nivolumab and ipilimumab will be fixed at FDA approved levels for each indication. Dosing of the drugs will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion is met. Patients who complete 12 months on study treatment and demonstrate clinical benefit with manageable toxicity will be given the opportunity to continue treatment for another 12 months upon agreement between investigator and drug manufacturers.

ELIGIBILITY:
Inclusion Criteria

1. Male or female ≥18 years old.
2. Patients with histologically confirmed unresectable Stage III or Stage IV metastatic melanoma who have not been previously treated with a CD24Fc, anti-CTLA4 and anti-PD1/PDL1 inhibitors with documented progression.
3. Measurable disease per RECIST v1.1 criteria using imaging scans, or peripheral lesions that can be adequately documented with a picture and a ruler even if they do not meet RECIST criteria.
4. Patients must have lesion accessible for sequential biopsy (core needle biopsy or excision preferred, fine needle aspiration not eligible).
5. ECOG performance status 0 or 1.
6. Women of child-bearing potential must have a negative serum pregnancy test within 24 hour of initiation of dosing and must agree to use an effective form of contraception during the study from the time of the negative pregnancy test up to 6 months after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraceptive in conjunction with a barrier method, or a double barrier method. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year. Fertile men must also agree to use an effective method of birth control while on study drug and up to 6 months after the last dose of study drug.
7. Patients must have fully recovered from the effects of any major surgery or significant traumatic injury within 14 days of C1D1.
8. Adequate hematologic, hepatic, and renal function, as defined below:

   * Absolute neutrophil count ≥1 X 109/L,
   * Hgb > 8 g/dL
   * Platelet count ≥ 75 X 109/L,
   * AST/ALT/bilirubin ≤3X ULN (patients with Gilbert syndrome can have higher bilirubin levels).
   * Creatinine ≤ 3 X ULN or calculated CrCl > 30 mL/min using Cockcroft- Gault formula.
9. Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements.

Exclusion Criteria

1. Active secondary malignancy, unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the Medical Monitor.
2. Investigational drug use within 28 days of C1D1.
3. Chemotherapy, targeted therapy, growth factors or radiation therapy within 14 days of C1D1.
4. Systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to C1D1.
5. Patients with known active CNS lesions are excluded (i.e., those with radiographically unstable, symptomatic lesions). However, patients treated with stereotactic therapy or surgery are eligible if they remain without clinical evidence of disease progression in the brain.
6. Has received a live vaccine within 28 days prior to C1D1.
7. A known active and clinically significant bacterial, fungal, or viral infection.
8. Active hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness, including patients who have an active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of combination of CD24Fc with Ipilimumab and Nivolumab | 4 weeks
  The rate of Grade 3 or above treatment-related adverse events (TRAE) at 4 weeks after first dosing of drugs.

SECONDARY OUTCOMES:
Profile of treatment related adverse events | 1 year
  To tabulate the treatment related adverse events in 1 year
The Objective Response Rate (OPR) | 1 year
  The rate of objective response with CD24Fc, Ipilimumab, Nivolumab combination therapy at 1 year
The Progression Free Survival (PFS) | 1 year
  The rate of Progression Free Survival with CD24Fc, Ipilimumab, Nivolumab combination therapy at 1 year.
The Overall Survival (OS) | 1 year
  The rate of Overall Survival with CD24Fc, Ipilimumab, Nivolumab combination therapy at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php